CLINICAL TRIAL: NCT02922335
Title: Effectiveness Trial of Treatment to Reduce Serious Antisocial Behavior in Emerging Adults With Mental Illness
Brief Title: Multisystemic Therapy-Emerging Adults Trial
Acronym: MST-EA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Oregon Social Learning Center (Other); Connecticut Department of Children and Families (Unknown); North American Family Institute (Unknown); Court Support Services Division (Unknown); Youth Villages (Other)
Responsible Party: Principal Investigator, Maryann Davis, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H0009053; 1R01MH108793-01 (NIH)
Record Dates: First submitted 2016-07-26; First posted 2016-10-04 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Antisocial Behavior
Keywords: Antisocial Behavior; Mental Illness; Emerging Adulthood; Criminal Behavior; Serious Mental Illness
MeSH Terms: conditions — Antisocial Personality Disorder; Mental Disorders; Criminal Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisystemic Therapy - Emerging Adults (Experimental): Multisystemic Therapy for Emerging Adults (MST-EA) is designed to help emerging adults (ages 18-21) with mental illness who have been in trouble with the law. MST-EA is a treatment program specifically for emerging adults, to increase skills and capacities that can help them reduce their antisocial behavior and help reduce problems caused by mental health illness, and alcohol or drug use when present.
  Interventions: Behavioral: Multisystemic Therapy for Emerging Adults
- Enhanced Treatment as Usual (Active Comparator): With Enhanced Treatment as Usual (E-TAU) emerging adults will get the treatments that they usually receive when they have a mental illness and have been in trouble with the law. They will receive travel vouchers for attending services, a card with an individualized list of contacts when in crisis, and facilitation with identifying need of services and accessing those services.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Multisystemic Therapy for Emerging Adults — MST-EA is a home-based therapy in which therapists work closely with each young adult. Therapists often also work with the young person's family, as appropriate. MST-EA is designed to help young people work on their own behavior. This treatment also involves the use of coaches who help young people develop skills for young adulthood.
  Other Names: Multisystemic Therapy for Transition-Age Youth (MST-TAY)
  Arms: Multisystemic Therapy - Emerging Adults
Behavioral: Enhanced Treatment as Usual — Standard services that a young person would receive if they have been in trouble with the law and also have a mental illness.
  Other Names: E-TAU
  Arms: Enhanced Treatment as Usual

SUMMARY:
This study's purpose is to test the effectiveness of a promising intervention for emerging adults (EAs) with mental illness (MI) and serious antisocial behavior in achieving the ultimate outcome of reduced antisocial behavior, and proximal intermediate outcomes. Multisystemic Therapy-Emerging Adults (MST-EA) is an adaptation of MST, a well-established, effective intervention for antisocial behavior in adolescents.

DETAILED DESCRIPTION:
Serious antisocial behavior, including criminal offending, is extremely costly to society. Rates of such behavior are highest during emerging adulthood. Antisocial behavior is especially high among emerging adults (EAs) with mental illness (MI); findings suggest the majority of EAs with MI will be arrested by age 25, most with multiple arrests, and for serious charges. Thus, there is a clear public health need for effective treatments to reduce serious antisocial behavior in EAs with MI. Astonishingly, there are no established interventions with evidence of efficacy to reduce serious antisocial behavior among EAs, with or without MI. Effective antisocial behavior interventions in adolescents address the comprehensive causes of that behavior. Similarly, this team has developed and completed research on a well-defined age-tailored intervention for EAs with MI and serious antisocial behavior that addresses the correlates of EA antisocial behavior, and provides MI treatment. The intervention is an adaptation of the well-established effective juvenile antisocial behavior intervention, Multisystemic Therapy (MST). MST-EA is a single source that targets the EA correlates of antisocial behavior, including gainful activity (school, work, housing, and positive relationships) and reduced substance use, in part by targeting the proximal mechanism of poor self-regulation. MST-EA also addresses these correlates through reducing MI symptoms. The investigative team has already established the safety, feasibility, and preliminary efficacy of this type of intervention in a successfully completed community-based open trial (R34MH081374-01, PI: Davis). The proposed study will rigorously evaluate the effectiveness of MST-EA for reducing serious antisocial behavior. Specifically, 240 EAs with MI and recent arrests or release from justice facilities will be randomized to receive MST-EA or Enhanced Treatment as Usual (E-TAU). Assessments will be completed at months 0, 2, 4, 6, 8, 12, and 16, with confirmation of outcome data using system records. The first aim will be to evaluate the effect over time of MST-EA for improving the ultimate outcome of treatment: reduced serious antisocial behavior. The second aim is to evaluate the effect of MST-EA on (a) the key proximal target of treatment (self-regulation) and (b) the proposed intermediate outcomes of treatment (gainful activity, substance use, and MI problems). The final aim will be to determine whether MST-EA's effect on the ultimate outcome is the result of its effect on the proximal target and intermediate outcomes of treatment. There is a current absence of any antisocial behavior treatments with demonstrated efficacy in this age group. The ultimate effect of the proposed research would be decreased antisocial behavior and other public health-related behaviors (MI symptoms, substance use, homelessness, unemployment) among one of the highest-risk populations of individuals with MI. With an emphasis on treatment mechanisms and the near absence of MI research focused on EAs, this innovative research has high potential to advance the field.

ELIGIBILITY:
Inclusion Criteria:

* age 16-26
* recent arrest or release from jail/prison/detention (within the past 18 months but excluding arrests for probation/parole violations)
* presence of mood, anxiety, and/or psychotic disorders
* able to reside in a stable community setting (not currently homeless, not currently inpatient; can include individual ready for discharge to the community)
* subject consent

Exclusion Criteria:

* actively psychotic, suicidal, or homicidal
* Pervasive Developmental Disorders (PDD) or mental retardation
* sex offending as the primary antisocial behavior
* adults unable to consent will also be excluded from this study

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 193 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in number and severity of criminal charges in official records in the 16 months pre-baseline compared with the 16 months post-baseline. | 16 months pre-baseline compared with 16 months post-baseline
  Changes from the Baseline in offending, measured in the number of offenses in the Self-Report Offending Scale, during the 16 months post-baseline.

SECONDARY OUTCOMES:
Changes from Baseline scores compared to 16 months post-Baseline Self-efficacy (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Self-efficacy measured using the General Self-Efficacy Scale (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Goal directness (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Goal directness measured using Wills Self Control Measures (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Responsibility taking (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Responsibility taking measured using sub-scale of the Behavioral Indicators of Conscientiousness (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Symptoms (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  The number and severity of symptoms measured using the Brief Symptom Inventory (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Treatment Usage (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  The number of hospitalizations, Emergency Room visits and treatment usage for psychiatric reasons (Self-Report and Archival records).
Changes from Baseline scores compared to 16 months post-Baseline Drug Screens (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  The number of positive drug screens from toxicology testing for tetrahydrocannabinol (THC), synthetic THC, amphetamines, methamphetamines, opiates, benzodiazepines, and cocaine.
Changes from Baseline scores compared to 16 months post-Baseline Substance Use and Problems(measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Frequency of substance use and substance-related problems reported on the Global Appraisal of Individual Needs (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Antisocial Peers (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Antisocial Peer Involvement measured using the Peer Delinquency Scale (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Interpersonal Competence (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Social Conflict and social functioning measured in the Interpersonal Competence Scale (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline Housing stability (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Housing stability as reported by participant and archival.
Changes from Baseline scores compared to 16 months post-Baseline Relationships (measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Network of Relationships Inventory (Self Report).
Changes from Baseline scores compared to 16 months post-Baseline School and Work(measured at 0,2,4,6,8,12 and 16 months). | Baseline to16 months
  Days in school or work measured as reported by participant and archival.

CONTACTS AND LOCATIONS:
Overall Officials: Maryann Davis, PhD, Principal Investigator — University of Massachusetts, Worcester; Ashli Sheidow, PhD, Principal Investigator — Oregon Social Learning Center
Locations (4):
- United States (4):
  - North American Family Institute, Hamden, Connecticut
  - North American Family Institute, Hartford, Connecticut
  - North American Family Institute, New Haven, Connecticut
  - Youth Villages, Johnson City, Tennessee

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sheidow AJ, McCart MR, Davis M. Multisystemic Therapy for Emerging Adults With Serious Mental Illness and Justice Involvement. Cogn Behav Pract. 2016 Aug;23(3):356-367. doi: 10.1016/j.cbpra.2015.09.003. PMID 28458504
- [Result] Davis M, Sheidow AJ, McCart MR. Reducing recidivism and symptoms in emerging adults with serious mental health conditions and justice system involvement. J Behav Health Serv Res. 2015 Apr;42(2):172-90. doi: 10.1007/s11414-014-9425-8. PMID 25023764